CLINICAL TRIAL: NCT00429988
Title: Ductal Lavage to Monitor and Treat High Risk Women
Brief Title: Study of Ductal Lavage in Women at High Risk for Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000378088; UCSF-TEMP01
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — In Situ Hybridization, Fluorescence; Polymerase Chain Reaction; Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Genetic: fluorescence in situ hybridization
Genetic: polymerase chain reaction
Genetic: proteomic profiling
Other: cytology specimen collection procedure
Other: immunohistochemistry staining method
Procedure: breast duct lavage

SUMMARY:
RATIONALE: Collecting samples of fluid using ductal lavage and nipple aspiration from participants at high risk for breast cancer to study in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This clinical trial is using ductal lavage to collect fluid from women at high risk for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the volume of atypical cells collected from ductal lavage in women at increased risk for breast cancer.

Secondary

* Determine assay techniques to analyze nipple aspirate fluid and ductal lavage fluid samples from these participants.
* Analyze the nipple aspirate fluid from these participants for specific and global protein signatures.
* Determine the replicability of markers in serial assays of these participants.
* Determine the percentage of participants with atypia on ductal lavage in which ductal lesions can be identified using ductoscopy.

OUTLINE: This is a multicenter study.

Participants undergo nipple aspirate fluid and ductal lavage fluid collection. Fluid samples are analyzed using cytological analysis, immunohistochemistry, fluorescent in situ hybridization, or in situ polymerase chain reaction. Protein patterns are identified using mass spectrometry.

Participants found to have atypia undergo repeat lavage at 3-6 months and 1 year. Participants with normal fluid samples undergo repeat lavage at 1 year.

PROJECTED ACCRUAL: A total of 30 participants will accrued for this study within 2-3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* High risk for breast cancer defined as 1 of the following:

  * History of atypical hyperplasia or atypia found on biopsy, fine-needle aspiration, or ductal lavage
  * Family history of cancer meeting at least 1 of the following criteria:

    * Single relative with multiple primary cancers
    * One or more relative under 40 years of age with breast cancer OR bilateral breast cancer
    * Two or more relatives with ovarian cancer
    * Two or more relatives with breast cancer and 1 is under 50 years of age
    * One or more relative with breast cancer plus ≥ 1 relative with ovarian cancer
    * Ashkenazi Jewish descent AND relative with breast cancer under 50 years of age OR ovarian cancer at any age
  * BRCA1 and/or BRCA2 mutation
  * Prior breast cancer in contralateral breast
  * Gail risk > 1.7%
  * Spontaneous nipple discharge
  * Serum estradiol > 10 pmol/L
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Over 18

Sex

* Female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Able to obtain breast duct fluids

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* More than 4 months since prior tamoxifen or raloxifene

Radiotherapy

* No prior radiotherapy to the breast

Surgery

* No prior incisional or excisional biopsy within 1.5 cm of nipple

Other

* No prior neoadjuvant therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women at increased risk for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2002-08; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Average number of atypical cells per ductal lavage sample

SECONDARY OUTCOMES:
Assay techniques development for nipple aspirate fluid and ductal lavage fluid analysis
Specific and global protein signature analysis of nipple aspirate
Replicability of markers in serial assays
Percentage of participants with atypia on ductal lavage in which ductal lesions can be identified using ductoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Laura J. Esserman, MD, MBA, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States